CLINICAL TRIAL: NCT00217360
Title: RCT to Evaluate the Effectiveness of a Targeted and Personalised Multifactorial Program to Reduce Further Falls and Injuries for Community-Dwelling Older Fallers Presenting to and Being Discharged Directly From an Emergency Department.
Brief Title: RCT to Reduce Further Falls and Injuries for Older Fallers Presenting to an Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Ageing Research Institute, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC 2001.034
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-09

CONDITIONS: Accidental Falls

INTERVENTIONS:
Behavioral: a customised multifactorial falls prevention program

SUMMARY:
This project is called "Falls Aren't Us" and aimed at evaluating the effectiveness of a customised falls prevention program for people aged 60 and over who were presented to the hospital Emergency Department following a fall and being discharged home. Recruitment for this randomized controlled trial has commenced in late December 2002 from several major public hospitals in the western, southern, and northern parts of Melbourne Metropolitan Region. Consented participants will receive a comprehensive falls risk assessment within one week of being discharged home from the Emergency Department and at twelve month following this initial assessment. Their falls risks will be monitored for twelve months through a falls diary. Following randomization, participants in the intervention group will receive a customised falls prevention program in addition to the usual care being put in place from the hospital Emergency Department.

DETAILED DESCRIPTION:
Older people presenting to an Emergency Department (ED) following a fall have high injury and hospitalisation rates. They are also at high risk of further falls and other adverse outcomes. However, there is currently limited available evidence to inform best practice.

The primary aim of this project is to evaluate the effectiveness of a targeted multi-factor intervention in improving health and well being of older people who present to an ED after a fall. It also aims to identify those within this high-risk population most likely to benefit from the intervention program.

Approximately 800 people aged 60 years and over will be invited to participate at the Emergency Department from the end of September 2002. Those who are eligible to participate will have a falls risk assessment in their own home and will be required to complete a falls diary for 12 months. There is a 50/50 chance (random allocation) that participants will receive an individualised falls prevention program.

The duration of a falls risk assessment is up to 2 hours and there is no cost involved. Participation in the research program will not affect routine management from the Emergency Department.

Becoming a participant may lessen the risk of having another fall and help others as well.

ELIGIBILITY:
Inclusion Criteria:

* presenting to the Emergency Department with the primary cause of presentation being a fall; aged 60 years or older;
* discharged directly home following emergency care; living in the community or a retirement village; willing to take part in the study;
* able to provide informed consent or has consent provided by a third party; able to comply with simple instructions;
* able to walk independently indoors with or without a gait aid.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2002-12; Study Completion 2006-12

PRIMARY OUTCOMES:
To evaluate the effectiveness of a customised multifactorial intervention in reducing falls and falls related injury rates, compared to "usual care".

SECONDARY OUTCOMES:
To accurately identify the circumstances, contributory factors and consequences of falls for older people presenting to Emergency Departments following a fall.
To evaluate the effectiveness of the intervention program in improving secondary health and well-being measures, including physical, psychological (fear of falling, depression), and quality of life indices.
To identify the physical, functional, and cognitive (executive function) parameters most strongly associated with good outcomeTo conduct an economic evaluation of the interventions and outcomes.
To provide guidelines for future management of high risk older people presenting to Emergency departments.

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Hill, PhD, Principal Investigator — National Ageing Research Institute
Locations (1):
- National Ageing Research Institute, Melbourne, Victoria, Australia